CLINICAL TRIAL: NCT04548232
Title: Shanghai Tenth People's Hospital，School of Medicine, Tongji University
Brief Title: Clinical Efficacy and Safety of a Laparoscopic Sleeve Gastrectomy in Obese Patients
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Qu, Professor, Shanghai 10th People's Hospital
Other Study IDs: LSG in Obese Patients
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Obesity
Keywords: Laparoscopic sleeve Gastrectomy; Nonalcoholic Fatty Liver; Type 2 Diabetes; Polycystic Ovary Syndrome; Acanthosis nigricans; Hyperuricemia; Hyperinsulinemia; Sleep apnea Syndrome
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Polycystic Ovary Syndrome; Acanthosis Nigricans; Hyperuricemia; Hyperinsulinism; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSG in obese: Patients with obesity underwent LSG. Divided into simple obese patients (without complications) and obese patients with complications
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Control group: healthy individuals with normal BMI

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — bariatric surgery
  Groups: LSG in obese

SUMMARY:
This study aim to evaluate the clinical efficacy and safety after laparoscopic sleeve gastrectomy in patients with obesity. 300 patients with obesity and 49 healthy individuals with normal BMI were enrolled.

DETAILED DESCRIPTION:
This study aim to evaluate the clinical efficacy and safety after laparoscopic sleeve gastrectomy in patients with obesity. 300 patients with obesity and 49 healthy individuals with normal BMI were enrolled.

All patients with obesity underwent LSG. A multidisciplinary team evaluated participants with obesity at baseline, 1, 3, 6, 12, 24, and 36 months after LSG. Anthropometrics, Metabolic indicators, sex hormones, menstruation，glucose-lipid metabolic markers, and hepatic steatosis assessed by FibroScan(CAP value and E value) were measured baseline and postoperative.

ELIGIBILITY:
Inclusion Criteria:

1) age ranged from 16~65 years old, 2) BMI over 37.5 kg/m2, or BMI over 32.5 kg/m2 with diabetes which meets the recommended cutoff for bariatric surgery of the Guidelines for surgical treatment of obesity accompanied with or without type 2 diabetes in China. -

Exclusion Criteria:

* 1) secondary cause of obesity such as hypothalamic obesity, Cushing syndrome, and hypophysis dysfunction, etc., 2) pregnancy or lactation, 3) contraindications for laparoscopic surgery, such as gastrointestinal diseases of intra-abdominal infection, adhesions, etc., 4) severe heart, liver and kidney dysfunction, 5) organic and systemic diseases intolerant of surgery.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 300 subjects with obesity or overweight
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis | 3 years
  hepatic steatosis assessed by FibroScan(CAP value and E value)

SECONDARY OUTCOMES:
BMI | 3 years
  BMI=weight(kg)/height(m)^2
Menstrual cycles | 3 years
  the total number of menstrual periods in the last year
Waist/hip Ratio | 3 years
  WHR=Waist Circumference in centimeter/Hip Circumference in centimeter
TT | 3 years
  total testosterone in nmol/L
FBG | 3 years
  fasting blood-glucose in mmol/L
PBG | 3 years
  postprandial blood-glucose in mmol/L
FINS | 3 years
  fasting serum insulin in mU/L
PINS | 3 years
  postprandial insulin in mU/L
ALT | 3 years
  alanine aminotransferase in U/L
AST | 3 years
  aspartate aminotransferase in U/L
UA | 3 years
  Uric acid in umol/L
HOMA-IR | 3 years
  Homeostatic model assessment insulin resistance index=FBG*FINS/22.5
HbA1c (%)， | 3 years
  Glycated hemoglobin
SHBG | 3 years
  sex hormone-binding globulin in nmol/L
FT | 3 years
  free testosterone (nmol/L)
DHEAS | 3 years
  Dehydroepiandrosterone Sulfate (ug/dl)
LDL-C | 3 years
  low-density lipoprotein cholesterol in mmol/L、
HDL-C | 3 years
  Hight-density lipoprotein cholesterol in mmol/L、
Fertility | 3 years
  sexual function, fertility

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Fang Y, Huang X, Du L, Ren H, Sheng C, Yang P, Huang Y, Qu S. Relationship of serum iron and thyroid hormone in obesity and after laparoscopic sleeve gastrectomy. BMC Endocr Disord. 2024 Nov 7;24(1):240. doi: 10.1186/s12902-024-01753-8. PMID 39511506
- [Derived] Ma B, Yang P, Gao J, Du L, Sheng C, Usman T, Wang X, Qu S. Relationship of Vitamin A and Thyroid Function in Individuals With Obesity and After Laparoscopic Sleeve Gastrectomy. Front Nutr. 2022 Mar 15;9:824193. doi: 10.3389/fnut.2022.824193. eCollection 2022. PMID 35399676